CLINICAL TRIAL: NCT00850590
Title: A Randomised, Placebo-controlled, Double-blind, Dose Escalation Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Doses of Rectal Suppositories Containing Between 5 and 15 mg NRL001 or Matching Placebo for Two Different Sized Suppositories (1 g and 2 g).
Brief Title: Study of Escalating Doses of NRL001 Given in Slow-release Rectal Suppositories of Different Weights
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: VP Clinical Development, Norgine Ltd
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NRL001-02/2008 (SUSD)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Experimental): NRL001 at 5, 7.5, and 10 mg administered in a dose escalating manner with placebo in a random position in the sequence. NRL001 is contained in either a 1 g or a 2 g slow release rectal suppository.
  Interventions: Drug: NRL001
- High Dose (Experimental): NRL001 at 10, 12.5, and 15 mg administered in a dose escalating manner with placebo in a random position in the sequence. NRL001 is contained in either a 1 g or a 2 g slow release rectal suppository.
  Interventions: Drug: NRL001

INTERVENTIONS:
Drug: NRL001 — Four single doses of NRL001 or placebo. NRL001 is administered at lower (5, 7.5 and 10 mg) or higher (10, 12.5 and 15 mg) doses in a slow release rectal suppository weighing either 1 g or 2 g.

SUMMARY:
Studies investigating single doses of different NRL001 formulations showed formulation-dependent differences in exposure, even though they had similar effects on mean anal resting pressure (MARP). This study is a first step in investigating the hypothesis that a better balance between desired anal effects and undesired systemic effects can be reached with a NRL001-slow release suppository than with previously studied formulations.

To this purpose, single doses of 5 to 15 mg, administered as 1 g and 2 g suppositories, are being investigated with regard to their pharmacokinetics and systemic effects (blood pressure, pulse rate, electrocardiographic heart rate).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers (as determined by medical history, physical examination, laboratory test values, vital signs, and electrocardiograms [ECGs] at screening) aged 18-45 years.
2. Non-smokers from 3 months of receiving first dose and for the duration of the study.
3. Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2.
4. Able and willing to receive rectal treatments.
5. Able to voluntarily provide written informed consent to participate in the study.
6. Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol.
7. Female volunteers must be postmenopausal (for at least one year and confirmed by serum FSH at screening), surgically sterile, practising true sexual abstinence, or use two highly effective methods of contraception as follows throughout the study until after post study physical: contraceptive implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), vasectomised partner or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository.
8. Hormonal and IUD methods of contraception must be established for a period of 3 months prior to dosing and cannot be changed or altered during the study.
9. Females of child bearing potential must have a negative pregnancy test at screening (β-HCG) and prior to each dosing.
10. Sexually active male volunteers must use condoms with their partners throughout the study and for 90 days after completion of the study in addition to their normal mode of contraception.
11. Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
12. Must be willing to consent to have data entered into The Over Volunteering Prevention System.
13. The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study.

Exclusion Criteria:

1. Positive for HIV, hepatitis B, or hepatitis C as demonstrated by the results of testing at screening.
2. History or presence of any significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
3. History or presence of aortic stenosis or hypertrophic cardiomyopathy.
4. History or presence of any ano-rectal conditions, clinically significant latex allergy or clinically significant drug allergy.
5. Presence of any ECG abnormalities (during rest or during the exercise stress test).
6. Pregnant or lactating females.
7. Laboratory values at screening which are >1.5x the upper limit of normal for that parameter or <1.5x the lower limit of normal for that parameter, as applicable, or which are abnormal or deemed to be clinically significant according to Bio-Kinetic Europe Ltds SOPs, unless agreed in advance by the Sponsor's Responsible Medical Officer and the Bio-Kinetic Investigator.
8. Current or history of drug or alcohol abuse or a positive drugs of abuse test at screening or check in.
9. Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.
10. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
11. Any significant illness during the screening period preceding entry into this study.
12. Donation of blood or blood products within 90 days prior to study drug administration, or at anytime during the study, except as required by this protocol.
13. Strenuous exercise during study conduct and one week prior to dosing (with the exception of the exercise stress test).
14. Consumption of alcoholic beverages within 24 hours prior to each dosing. Abstinence is required during study confinement.
15. Consumption of xanthine-containing products within 24 hours of each dosing and during study confinement.
16. Use of any disallowed concomitant medication including over-the-counter items within 14 days prior to study drug administration until the end of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of different strengths of NRL001 rectal suppositories | Up to 36 hours post-dose

SECONDARY OUTCOMES:
Dose-related effects on cardiovascular parameters compared with placebo. | Up to 36 hours post-dose
To assess the safety and tolerability of NRL001. | Up to 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; David Bell, MRCGP MFPM, Principal Investigator — Biokinetic Europe Ltd
Locations (1):
- Bio-Kinetic Europe Limited, Belfast, United Kingdom

REFERENCES:
- [Derived] Bell D, Pediconi C, Jacobs A. Randomised clinical trial: study of escalating doses of NRL001 given in rectal suppositories of different weights. Colorectal Dis. 2014 Mar;16 Suppl 1:16-26. doi: 10.1111/codi.12542. PMID 24499493